CLINICAL TRIAL: NCT04378088
Title: The Colon Endoscopic Bubble Scale (CEBuS); Validation Study
Acronym: CEBuS
Status: Completed | Type: Observational
Sponsor: Portuguese Oncology Institute, Coimbra (Other)
Responsible Party: Principal Investigator, Filipe Taveira, Principal Investigator, Portuguese Oncology Institute, Coimbra
Other Study IDs: PortugueseOIC 005
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Colon Polyp
Keywords: Colonoscopy; Quality; Bowel; Preparation
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 - experts: Evaluation of 15 images for each of the proposed 3 grade scale (45 images in total), randomly distributed to validate de scale; images will be assessed twice by the participants with a two-week interval in both study phases (the random distribution will vary between both evaluations).
  Together with the assessment of each image the participant is invited to choose one of possible three clinical actions (do nothing, wash with water and wash with simethicone)
  Interventions: Other: Validation of CEBuS
- Group 2 - mix experts/trainee: If intra and interobserver rates in group 1 are >0.7 proceed to group 2 evaluation with the same intervention.
  Evaluation of 15 images for each of the proposed 3 grade scale (45 images in total), randomly distributed to validate de scale; images will be assessed twice by the participants with a two-week interval in both study phases (the random distribution will vary between both evaluations).
  Together with the assessment of each image the participant is invited to choose one of possible three clinical actions (do nothing, wash with water and wash with simethicone)
  Interventions: Other: Validation of CEBuS

INTERVENTIONS:
Other: Validation of CEBuS — Validation of a new score for bubbles in the colon.

SUMMARY:
Colonoscopy is currently accepted as the gold standard in screening, surveillance and prevention for colorectal cancer (CRC), and therefore, its quality is a major priority.

The quality of colonoscopy is greatly dependent on the quality of the bowel preparation, which can be limited by stool, foam, bubbles and other debris. In fact, colonic bubbles are described in 30 to 40% of colonoscopies, possibly undermining the quality of the exam, impairing the endoscopists view, demanding the further use of water or simethicone and eventually increasing fatigue and costs, while diminishing diagnostic accuracy.

Although previous attempts, to date no endoscopic scale is validated regarding the presence of bubbles and most widely accepted and already validated scales do not include the presence or absence of bubbles in their definition, leading to the use of different home-made scales in randomized trials and impairing any solid meta-analysis conclusion. As so, the goal of this study is to develop and validate a new colonic bubble score (Colon Endoscopic Bubble Scale - CEBuS).

DETAILED DESCRIPTION:
Colonoscopy bowel preparation quality is a major concern since inadequate bowel preparation can reach levels as high as 30% which lead to several guidelines in this area, with the recent recommendation of at least 90% of good bowel preparations for all colonoscopies. In fact colonic mucosal visualization can be limited by residual stool, bubbles, bile and other debris increasing the risk of missing lesions.

Around 30 to 40% of the exams can have bubbles increasing the risk of missing lesions and in the other hand increasing the time of the exam, generating more fatigue in the endoscopist and increasing the costs.

The influence of colon bubbles in bowel preparation and strategies to solve them, for example with the use of simethicone in the bowel preparation, were addresses in recent studies, summarized in a 2018 meta-analysis recommending the use of simethicone in the bowel preparation scheme.

Current recommendations advise the use of validated scales to evaluate bowel preparation quality, but the three major validated scales, Boston, Ottawa and Aronchick, does not address the problem of graduation of colonic bubbles and possible actions to undertake regarding the severity of the bubbles concentration. The advent of multiple randomized trials addressing the use of simethicone in the bowel preparation to reduce or eliminate bubble formation lead to attempts to design scales to graduate the concentration of bubbles in the colon.

To date suggested scales are heterogeneous regarding the graduation (3 to 4 levels), defining criteria for each level with some based on percentage of colonic circumference obscured by bubbles to the amount of bubbles that could lead to miss a polyp of 5 or 10 millimetres.Two recently published studies on the influence of simethicone on bowel preparation tried to validate a colonic bubble scale, based on previous suggested and non-validated scales, although with only fair to moderate inter-observer variability.

Therefore, the main goal of this project is to build and validate a comprehensive scale to graduate bubbles in the colon, assessing the inter- and intra-observer reliability of the scale. As a secondary objective, to determine the clinical attitude more frequent for each grade of the bubbles scale, among experts and residents.

Aims: Build and validate a new colonic bubble score (Colon Endoscopic Bubble Scale - CEBuS).

ELIGIBILITY:
Inclusion Criteria:

* For the expert group: at least 15 years of regular practice in colonoscopy
* For the trainee group: 5 years or less in the practice of colonoscopy

Exclusion Criteria:

* Non endoscopist and if out of the experience standards required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Were selected for the study 23 observers - 10 experts and 13 in-training/young specialists endoscopists from six European countries (Portugal, France, Italy, Romania, Poland and Slovakia).
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Reliability and reproducibility validation of the Colon Endoscopic Bubble Scale (CEBuS) | 1 month
  Evaluate the Intraclass correlation coefficients (ICC) and Fleiss kappa test
  The Colon Endoscopic Bubble Scale (CEBuS) was designed with a 3 grades scale:
  CEBuS-0 - no or minimal amount of bubbles, covering less than 5% of the surface, not relevant for adequate mucosa visibility (better outcome) CEBuS-1 - moderate amount of bubbles, covering between 5% and 50% of the surface, affecting mucosa visibility and requiring additional time for removal CEBuS-2 - severe amount of bubbles, covering more than 50% of the surface, obscuring mucosa visibility and requiring additional time for removal (worse outcome)

SECONDARY OUTCOMES:
Evaluation of the clinical attitude | 1 month
  Evaluated by the Intraclass correlation coefficients (ICC) and Fleiss kappa test
Influence of experience in the Colon Endoscopic Bubble Scale (CEBuS) | 1 month
  Evaluated by the Intraclass correlation coefficients (ICC) and Fleiss kappa test
  The Colon Endoscopic Bubble Scale (CEBuS) was designed with a 3 grades scale:
  CEBuS-0 - no or minimal amount of bubbles, covering less than 5% of the surface, not relevant for adequate mucosa visibility (better outcome) CEBuS-1 - moderate amount of bubbles, covering between 5% and 50% of the surface, affecting mucosa visibility and requiring additional time for removal CEBuS-2 - severe amount of bubbles, covering more than 50% of the surface, obscuring mucosa visibility and requiring additional time for removal (worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Filipe Taveira, MD, Principal Investigator — Gastroenterology Department of Portuguese Oncology Institute of Coimbra
Locations (1):
- Portuguese Oncology Institute - Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hassan C, Fuccio L, Bruno M, Pagano N, Spada C, Carrara S, Giordanino C, Rondonotti E, Curcio G, Dulbecco P, Fabbri C, Della Casa D, Maiero S, Simone A, Iacopini F, Feliciangeli G, Manes G, Rinaldi A, Zullo A, Rogai F, Repici A. A predictive model identifies patients most likely to have inadequate bowel preparation for colonoscopy. Clin Gastroenterol Hepatol. 2012 May;10(5):501-6. doi: 10.1016/j.cgh.2011.12.037. Epub 2012 Jan 10. PMID 22239959
- [Background] Kaminski MF, Thomas-Gibson S, Bugajski M, Bretthauer M, Rees CJ, Dekker E, Hoff G, Jover R, Suchanek S, Ferlitsch M, Anderson J, Roesch T, Hultcranz R, Racz I, Kuipers EJ, Garborg K, East JE, Rupinski M, Seip B, Bennett C, Senore C, Minozzi S, Bisschops R, Domagk D, Valori R, Spada C, Hassan C, Dinis-Ribeiro M, Rutter MD. Performance measures for lower gastrointestinal endoscopy: a European Society of Gastrointestinal Endoscopy (ESGE) Quality Improvement Initiative. Endoscopy. 2017 Apr;49(4):378-397. doi: 10.1055/s-0043-103411. Epub 2017 Mar 7. PMID 28268235
- [Background] Yoo IK, Jeen YT, Kang SH, Lee JH, Kim SH, Lee JM, Choi HS, Kim ES, Keum B, Chun HJ, Lee HS, Kim CD. Improving of bowel cleansing effect for polyethylene glycol with ascorbic acid using simethicone: A randomized controlled trial. Medicine (Baltimore). 2016 Jul;95(28):e4163. doi: 10.1097/MD.0000000000004163. PMID 27428209
- [Background] Matro R, Tupchong K, Daskalakis C, Gordon V, Katz L, Kastenberg D. The effect on colon visualization during colonoscopy of the addition of simethicone to polyethylene glycol-electrolyte solution: a randomized single-blind study. Clin Transl Gastroenterol. 2012 Nov 29;3(11):e26. doi: 10.1038/ctg.2012.16. PMID 23238113
- [Background] Pan P, Zhao SB, Li BH, Meng QQ, Yao J, Wang D, Li ZS, Bai Y. Effect of supplemental simethicone for bowel preparation on adenoma detection during colonoscopy: A meta-analysis of randomized controlled trials. J Gastroenterol Hepatol. 2019 Feb;34(2):314-320. doi: 10.1111/jgh.14401. Epub 2018 Aug 27. PMID 30069899
- [Background] Calderwood AH, Jacobson BC. Comprehensive validation of the Boston Bowel Preparation Scale. Gastrointest Endosc. 2010 Oct;72(4):686-92. doi: 10.1016/j.gie.2010.06.068. PMID 20883845
- [Background] Rostom A, Jolicoeur E. Validation of a new scale for the assessment of bowel preparation quality. Gastrointest Endosc. 2004 Apr;59(4):482-6. doi: 10.1016/s0016-5107(03)02875-x. PMID 15044882
- [Background] Aronchick CA, Lipshutz WH, Wright SH, Dufrayne F, Bergman G. A novel tableted purgative for colonoscopic preparation: efficacy and safety comparisons with Colyte and Fleet Phospho-Soda. Gastrointest Endosc. 2000 Sep;52(3):346-52. doi: 10.1067/mge.2000.108480. PMID 10968848
- [Background] Spada C, Cesaro P, Bazzoli F, Saracco GM, Cipolletta L, Buri L, Crosta C, Petruzziello L, Ceroni L, Fuccio L, Giordanino C, Elia C, Rotondano G, Bianco MA, Simeth C, Consalvo D, De Roberto G, Fiori G, Campanale M, Costamagna G. Evaluation of Clensia(R), a new low-volume PEG bowel preparation in colonoscopy: Multicentre randomized controlled trial versus 4L PEG. Dig Liver Dis. 2017 Jun;49(6):651-656. doi: 10.1016/j.dld.2017.01.167. Epub 2017 Feb 3. PMID 28233684
- [Background] Repici A, Cestari R, Annese V, Biscaglia G, Vitetta E, Minelli L, Trallori G, Orselli S, Andriulli A, Hassan C. Randomised clinical trial: low-volume bowel preparation for colonoscopy - a comparison between two different PEG-based formulations. Aliment Pharmacol Ther. 2012 Oct;36(8):717-24. doi: 10.1111/apt.12026. Epub 2012 Aug 28. PMID 22924336
- [Background] Guo R, Wang YJ, Liu M, Ge J, Zhang LY, Ma L, Huang WY, Zhai HH. The effect of quality of segmental bowel preparation on adenoma detection rate. BMC Gastroenterol. 2019 Jul 8;19(1):119. doi: 10.1186/s12876-019-1019-8. PMID 31286888
- [Background] Zhang S, Zheng D, Wang J, Wu J, Lei P, Luo Q, Wang L, Zhang B, Wang H, Cui Y, Chen M. Simethicone improves bowel cleansing with low-volume polyethylene glycol: a multicenter randomized trial. Endoscopy. 2018 Apr;50(4):412-422. doi: 10.1055/s-0043-121337. Epub 2017 Nov 13. PMID 29132175
- [Background] Rishi M, Kaur J, Ulanja M, Manasewitsch N, Svendsen M, Abdalla A, Vemala S, Kewanyama J, Singh K, Singh N, Gullapalli N, Osgard E. Randomized, double-blinded, placebo-controlled trial evaluating simethicone pretreatment with bowel preparation during colonoscopy. World J Gastrointest Endosc. 2019 Jun 16;11(6):413-423. doi: 10.4253/wjge.v11.i6.413. PMID 31236194
- [Background] Moraveji S, Casner N, Bashashati M, Garcia C, Dwivedi A, Zuckerman MJ, Carrion A, Ladd AM. The role of oral simethicone on the adenoma detection rate and other quality indicators of screening colonoscopy: a randomized, controlled, observer-blinded clinical trial. Gastrointest Endosc. 2019 Jul;90(1):141-149. doi: 10.1016/j.gie.2019.03.018. Epub 2019 Mar 26. PMID 30926430